CLINICAL TRIAL: NCT04594395
Title: Defining the COVID-19 Immunity Denominator in the Mekong: a Cross-Sectional Seroprevalence Study of SARS-CoV-2 in Healthy Volunteers
Brief Title: Defining the COVID-19 Immunity Denominator in the Mekong: a Cross-Sectional Seroprevalence Study of SARS-CoV-2 in HealthyVolunteers
Status: Withdrawn | Type: Observational
Why Stopped: Study never initiated in Cambodia
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000083; 000083-I
Record Dates: First submitted 2020-10-17; First posted 2020-10-20 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-10

CONDITIONS: Healthy Volunteers
Keywords: Mobile Units; SARS-CoV-2 Immunoglobulin-Positive; Antibody-Based Tests; ELISA; Phnom Penh

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood, serum

GROUPS / COHORTS (2):
- Healthy volunteers: Any adult aged 18 to 65 years of age living in Phnom Penh that is sufficiently healthy and willing to undergo fingerstick by the mobile unit for SARS-CoV-2 ELISA assays.
- Household contacts: Adult relatives of the healthy volunteers.

SUMMARY:
Background:

In early 2020, many people thought Cambodia would have a serious COVID-19 outbreak due to the high number of Chinese travelers going to Cambodia. But as of June 14, 2020, only 128 cases of COVID-19 have been identified in the country. Many of these cases have been from people who had traveled in Europe. Researchers want to do antibody tests on blood from a sampling of people in Phnom Penh to learn the infection risks for people in the greater Phnom Penh area.

Objective:

To estimate the level of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) in the blood of people living in Phnom Penh, Cambodia.

Eligibility:

Healthy males and females age 18-65 living in Phnom Penh since January 2020.

Design:

A mobile unit will travel to schools, shopping areas, parks, and pagodas around Phnom Penh.

Participants will be screened with questions about their age and where they live. They will have blood taken via fingerstick. About 80 uL of blood will be taken. It will be tested for SARS-CoV-2. This visit will take about 30 minutes.

If the test result is positive, participants will be contacted by phone. They will be asked to have a second blood draw. This time, 20 mL of blood will be taken. They can have this visit at their home or in a clinic. This visit will take about 30 minutes.

If a participant has an adverse event, the mobile units and at-home units will have the tools needed to aid the participant. If needed, the participant will be sent to a nearby clinic.

DETAILED DESCRIPTION:
This is a cross-sectional study performed annually over 3 years to procure blood samples by fingerstick from healthy individuals living in the Phnom Penh area to evaluate seroprevalence to SARS-CoV-2. A mobile unit will move between various markets, schools, hospitals, clinics, parks, and other public places with local authority permissions. Participants with a positive result on the screening SARS-CoV-2 ELISA will be contacted via telephone (since there is not reliable mail in Cambodia) and invited to undergo an additional blood draw via venipuncture during a home visit by the mobile team within 180 days of the initial sample collection. This visit may also be conducted by CCDC/CNM/MOH study staff at a local clinic. Up to 10 of their adult household contacts will be invited to enroll and screen at this time via fingerstick for SARS-CoV-2 ELISA as part of an enriched sampling scheme to boost the probability of identifying SARSCoV- 2 immune individuals; those with positive results will be invited to undergo follow-up venipuncture as described above. Venipuncture samples will be used to study the immune responses of Cambodians to the novel coronavirus.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Stated willingness to comply with all study procedures and availability for the duration of the study.
2. Male or female, aged 18 - 65 years of age.
3. Residing in Phnom Penh since January 1, 2020.
4. Ability to provide consent.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Any acute illness requiring a visit to a clinic or hospital on the same day as study enrollment.
2. Any underlying, chronic, or current medical condition that, in the opinion of the investigator, would interfere with participation in the study (e.g., inability or great difficulty in drawing blood).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Advertising and recruitment in this province will mainly be via word of mouth using health staff and the local village chiefs to communicate to the general public when and where the mobile unit will be sampling. Large signs and banners will be made to hang wherever the mobile unit set up in the designated area. We anticipate having to screen no more than 2,500 individuals per year to enroll our target of 2,000 participants per year over the next 3 years. We have no pre-set male:female ratios or age structures. We do plan to sample many different small clusters from the majority of Phnom Penh s administrative districts. Up to 200 household contacts may also be enrolled each year, bringing the overall total to 2,200 individuals enrolled per year. To account for screen failures, our total accrual ceiling over 3 years is 8,100.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-09-24 (Actual); Primary Completion 2021-09-24 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Presence or absence of SARSCoV-2 immunoglobulin in participant sera by ELISA optical density change. | Enrollment Day 1 (and Study Visit 2 if applicable)
  Using convenience sampling at randomized points across Phnom Penh, ELISAs to the SARS-CoV-2 full-length spike and ribonucleocapsid protein (RNP) antigens will be used as these are the most sensitive and specific to be interpreted in the setting of any background noise introduced by Cambodian sera, and because they are less expensive and amenable to high-throughput processing.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica E Manning, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (2):
- Cambodia (2):
  - Cambodian Center for Communicable Disease (CCDC), Ministry of Health (MOH), Phnom Penh
  - National Malaria Center (CNM), Ministry of Health (MOH), Phnom Penh

REFERENCES:
- [Background] Lang Z, Reiczigel J. Confidence limits for prevalence of disease adjusted for estimated sensitivity and specificity. Prev Vet Med. 2014 Jan 1;113(1):13-22. doi: 10.1016/j.prevetmed.2013.09.015. PMID 24416798